CLINICAL TRIAL: NCT07146009
Title: Targeted Nerve Surgery for the Prevention of Post-Mastectomy Pain Syndrome: A Randomized Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Reconstructive Surgery Alliance (Other Government)
Responsible Party: Principal Investigator, Kari Colen, Medical Doctor, Advanced Reconstructive Surgery Alliance
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R-2025.02.25.01
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Post-mastectomy pain syndrome (PMPS); Breast reconstruction; Regenerative Peripheral Nerve Interfaces; Targeted Muscle Reinnervation
MeSH Terms: conditions — Breast Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Patients receiving standard medical therapies for PMPS prevention (e.g., pharmacologic pain management, physical therapy).
  Interventions: Other: Standard of Care (Investigator Choice)
- Nerve Surgery (Experimental): Patients undergoing prophylactic nerve surgery (RPNI) during second-stage implant exchange after tissue expander based breast reconstruction.
  Interventions: Procedure: Nerve Surgery

INTERVENTIONS:
Procedure: Nerve Surgery — Patients undergoing prophylactic nerve surgery (RPNI) during second-stage implant exchange after tissue expander based breast reconstruction.
  Arms: Nerve Surgery
Other: Standard of Care (Investigator Choice) — Patients receiving standard medical therapies for PMPS prevention (e.g., pharmacologic pain management, physical therapy).
  Arms: Standard of care

SUMMARY:
Post-Mastectomy Pain Syndrome (PMPS) is a chronic pain condition often caused by neuroma formation and nerve injury following breast cancer surgery. Standard breast reconstruction protocols typically do not address damaged intercostal nerves, leaving patients at risk for persistent nerve-related pain.

Prophylactic nerve surgery techniques, such as Targeted Muscle Reinnervation (TMR) and Regenerative Peripheral Nerve Interfaces (RPNI), offer innovative approaches to prevent neuroma formation by managing damaged nerves during surgery. This study will evaluate whether incorporating prophylactic nerve surgery during second-stage implant exchange after tissue expander based breast reconstruction can reduce the incidence of PMPS compared to standard medical therapies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) undergoing second-stage implant exchange as part of tissue expander based breast reconstruction.
* Patients with no prior diagnosis of PMPS.

Exclusion Criteria:

* Prior nerve surgery in the chest region or chronic pain conditions unrelated to mastectomy.
* Recent chest radiation (<6 months), severe scarring, or active infection.
* Uncontrolled diabetes, high-dose corticosteroids, or immunosuppressive therapy.
* Psychiatric or cognitive impairments.
* Pregnancy, or active lactation.
* Autologous tissue based breast reconstruction.
* Participation in another study within 6 months or inability to comply with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-02-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post-Mastectomy Pain Syndrome | Pre-operative visit (baseline) to 12 months.
  Incidence of PMPS, defined as persistent pain beyond 6 months postoperatively.

SECONDARY OUTCOMES:
Breast Cancer Pain Questionnaire | Pre-operative visit (baseline) to 12 months.
  Pain severity scores at 3, 6, and 12 months.
Adverse event rates | Pre-operative visit (baseline) to 12 months.
  Complication and adverse event rates.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Colen, MD, Principal Investigator — Advanced Reconstructive Surgery Alliance

IPD SHARING:
Plan to Share IPD: No